CLINICAL TRIAL: NCT04393402
Title: Lung Ultrasound Score in Covid 19 Infectious Disease in Critical Care
Brief Title: Lung Ultrasound Score in Covid 19 Infectious Disease in Critical Care (LUS-COVID19)
Acronym: LUS-COVID19
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 20reamedcovid03
Record Dates: First submitted 2020-05-15; First posted 2020-05-19 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: COVID

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Covid-19 and admitted in critical care unit
  Interventions: Procedure: lung ultrasound (LUS)

INTERVENTIONS:
Procedure: lung ultrasound (LUS) — Patients with Covid-19 Disease and admitted in critical care unit will be performed a LUS

SUMMARY:
It might be necessary with Sars-Cov2 pneumopathy patient to repeat thoracic images, the tomodensitometry ones in particular. This task is difficult and nearly impossible for several reasons: respiratory and hemodynamic unstable patient, prone position and due to the high contagious nature of the disease.

The lung ultrasound is an easy tool, fast (between 5 and 10 minutes) and as a limited training.

In the context of the Sars-Cov2 epidemic, Buonsenso and al case report depict the first lung ultrasound for a Covid 19 patient.

Peng and al in Intensive Care Medicine accentuate the usefulness of this particular technic.

In the American Journal of Respiratory and Critical Care Medicine, a study has been published as a point-of-care, in which the doctors reported using the lung ultrasound with intensive and critical care patient.

In Critical Care 2016, it has been showed that ultrasound allowed with neat precisions, to predict severe ARDS patient response to the prone position, all-cause.

Another researchers team found a good correlation between lung ultrasound, the SOFA, APACHE II, CPIS score, and patient mortality.

And a new applicability in the pulmonary recruitment by PEEP titration has been presented.

The aim of this study is to evaluate the lung ultrasound in Covid19 ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Sars-Cov2 patient, with PCR method qualitative or quantitative as usual.
* Intensive or critical care admission
* ARDS with PaO2/FiO2 <300 at the admission
* Ventilatory support or oxygen-therapy

Exclusion Criteria:

* Age < 18 years-old
* Pregnancy
* Patient with tutor- or curatorship or in prison

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with diagnose of Covid 19 by usully method, and admitted in critical care unit for oxygen-therapy or ventilatory support.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
LUS applicability with COVID 19 | 10 months
  In dorsal position, or in prone position, the two hemithorax will be subdivided in 6 parts, and a score will be attributed with the following criteria : A-Lines (0 point), > 3 B-lines (1 point), B-Lines coalscent (2 points), and pulmonary consolidation (3 points). For the echography we can use a convexe sonde, or a "cardiac" sonde.

SECONDARY OUTCOMES:
Radiographic correlation (chest Xray and tomodensitometry) | 10 months
  Comparison between Xray / CT scan exam and LUS
LUS Mortality prediction | 10 months
  according to LUS score, ventilatory mode and parameters, medical history and bood analysis results
Prediction of Prone position response | 10 months
  comparison of LUS score depending of the position used for performing LUS

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No
No data sharing plan has been established